CLINICAL TRIAL: NCT04602325
Title: Systemic Biomarkers of Brain Injury From Hyperammonemia
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Nicholas Ah Mew, MD, Children's National Research Institute
Other Study IDs: 14021; R21TR003166-01 (NIH)
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Urea Cycle Disorder; Organic Acidemia; Maple Syrup Urine Disease; Glutaric Acidemia I; Fatty Acid Oxidation Disorder; Hypoxic-Ischemic Encephalopathy
Keywords: N-acetylglutamate Synthetase Deficiency; Carbamyl Phosphate Synthetase Deficiency; Ornithine Transcarbamylase Deficiency; Argininosuccinate Synthetase Deficiency; Argininosuccinate Lyase Deficiency; Arginase Deficiency; Hyperammonemia-Hyperornithinemia-Homocitrullinuria; Medium Chain-Acyl CoA Dehydrogenase Deficiency; Very Long Chain-Acyl CoA Dehydrogenase Deficiency; Trifunctional Protein Deficiency; Long Chain Hydroxyacyl-CoA Dehydrogenase Deficiency; Carnitine Palmitoyltransferase I or II Deficiency; Carnitine/Acylcarnitine Translocase Deficiency; Primary Carnitine Transport Deficiency
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Maple Syrup Urine Disease; Glutaric Acidemia I; Hypoxia-Ischemia, Brain; N-acetyl glutamate synthetase deficiency; Carbamoyl-Phosphate Synthase I Deficiency Disease; Ornithine Carbamoyltransferase Deficiency Disease; Citrullinemia; Argininosuccinic Aciduria; Hyperargininemia; HHH syndrome; Medium chain acyl CoA dehydrogenase deficiency; VLCAD deficiency; Trifunctional Protein Deficiency With Myopathy And Neuropathy; Carnitine-Acylcarnitine Translocase Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Discarded blood samples will be obtained from such laboratory tests in order to measure S100B, NSE, and UCHL1 levels at baseline (normal blood ammonia), which will provide data on biomarker levels following recovery from a hyperammonemic episode.
  During hospitalization for metabolic decompensation or for hypoxic-ischemic encephalopathy, sequential measurements of S100B, NSE and UCHL1 levels will be obtained from discarded blood samples.
  S100B, NSE, and UCHL1 levels will again be obtained from collected discarded blood samples at all subjects' next outpatient visit following their hospitalization, to determine if levels return to baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Inherited Hyperammonemias: A clinical diagnosis of 1 of 7 diagnosed urea cycle disorders:
  1. N-acetylglutamate Synthetase Deficiency (NAGS)
  2. Carbamyl Phosphate Synthetase Deficiency (CPSD)
  3. Ornithine Transcarbamylase Deficiency (OTCD)
  4. Argininosuccinate Synthetase Deficiency (ASD)
  5. Argininosuccinate Lyase Deficiency (ALD)
  6. Arginase Deficiency (AD)
  7. Hyperammonemia-Hyperornithinemia-Homocitrullinuria (HHH)
  A clinical diagnosis of 1 of 2 organic acidemias:
  1. Propionic Acidemia (PA)
  2. Methylmalonic Acidemia (MMA)
- Acute Metabolic Disorder + Neurological Sequelae: Acute metabolic disorder without hyperammonemia but with neurological sequelae:
  1. Maple Syrup Urine Disease (MSUD)
  2. Glutaric Acidemia (GA1)
- Fatty Acid Oxidation Disorders: Acute metabolic disorder without hyperammonemia and without neurological sequelae:
  1. Medium Chain-Acyl CoA Dehydrogenase Deficiency
  2. Very Long Chain-Acyl CoA Dehydrogenase Deficiency
  3. Trifunctional Protein Deficiency
  4. Long Chain Hydroxyacyl-CoA Dehydrogenase Deficiency
  5. Carnitine Palmitoyltransferase I or II Deficiency
  6. Carnitine/Acylcarnitine Translocase Deficiency
  7. Primary Carnitine Transport Deficiency
- Hypoxic-Ischemic Encephalopathy: Patients with hypoxic-ischemic encephalopathy

SUMMARY:
Ammonia is a waste product of protein and amino acid catabolism and is also a potent neurotoxin. High blood ammonia levels on the brain can manifest as cytotoxic brain edema and vascular compromise leading to intellectual and developmental disabilities. The following aims are proposed:

Aim 1 of this study will be to determine the chronology of biomarkers of brain injury in response to a hyperammonemic (HA) brain insult in patients with an inherited hyperammonemic disorder.

Aim 2 will be to determine if S100B, NSE, and UCHL1 are altered in patients with two other inborn errors of metabolism, Maple Syrup Urine Disease (MSUD) and Glutaric Acidemia (GA1).

DETAILED DESCRIPTION:
Ammonia is a waste product of protein and amino acid catabolism and is also a potent neurotoxin. The onslaught of high blood ammonia levels on the brain can manifest as cytotoxic brain edema and vascular compromise leading to intellectual and developmental disabilities. In addition, clinical hyperammonemia recurs at varying intervals, which can increase the cumulative damage to the brain and the chance of irreversible coma and death during a hyperammonemia episode due to vascular compromise or brain herniation. The threshold of tolerance for elevated blood ammonia is very low and concentrations above 100 µM can cause brain dysfunction manifested as nausea, vomiting, lethargy, and abnormal behavior; higher concentrations can cause coma and even death. Failure to remove ammonia can be due to inherited defects of the urea cycle, some defects in amino acid catabolism, and degradation of fatty acids.

Aim 1 - To determine the chronology of biomarkers of brain injury - S100B, NSE, and UCHL1 - in response to a hyperammonemic (HA) brain insult in patients with an inherited hyperammonemic disorder. We hypothesized that elevations of S100B, NSE, and UCHL1 will parallel the rise in blood ammonia. These biomarkers will be measured concurrently to ammonia levels throughout hospitalizations for HA until normalization of patient's blood ammonia and mental status.

Aim 2 - To determine if S100B, NSE, and UCHL1 are altered in patients with two other inborn errors of metabolism in which the primary pathology is neurological injury, Maple Syrup Urine Disease (MSUD) and Glutaric Acidemia (GA1). We hypothesize that neuronal and astroglial injury in these disorders may also result in increased levels of S100B, NSE, and UCHL1.

Metabolic patients will be enrolled either during a hospitalization or in outpatient clinic, but outpatient enrollment is preferred. Metabolic patients typically have multiple laboratory tests performed at their outpatient visits. We will obtain the discarded blood samples from such laboratory tests in order to measure S100B, NSE, and UCHL1 levels at baseline (normal blood ammonia), which will provide data on biomarker levels following recovery from a hyperammonemic episode.

During hospitalization for metabolic decompensation or for hypoxic-ischemic encephalopathy, sequential measurements of S100B, NSE and UCHL1 levels will be obtained from discarded blood samples. We will obtain S100B, NSE, and UCHL1 levels from collected discarded blood samples at all subjects' next outpatient visit following their hospitalization, to determine if levels return to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Inherited Hyperammonemias:

   1. A clinical diagnosis of 1 of 7 diagnosed urea cycle disorders:

      * N-acetylglutamate Synthetase Deficiency (NAGS)
      * Carbamyl Phosphate Synthetase Deficiency (CPSD)
      * Ornithine Transcarbamylase Deficiency (OTCD)
      * Argininosuccinate Synthetase Deficiency (ASD)
      * Argininosuccinate Lyase Deficiency (ALD)
      * Arginase Deficiency (AD)
      * Hyperammonemia-Hyperornithinemia-Homocitrullinuria (HHH)
   2. A clinical diagnosis of 1 of 2 organic acidemias:

      * Propionic Acidemia (PA)
      * Methylmalonic Acidemia (MMA)
2. Acute metabolic disorder without hyperammonemia, with neurological sequelae

   1. Maple Syrup Urine Disease (MSUD)
   2. Glutaric Acidemia (GA1)
3. Acute metabolic disorder without hyperammonemia and without neurological sequelae

   * Fatty Acid Oxidation Disorders:
   * Medium Chain-Acyl CoA Dehydrogenase Deficiency
   * Very Long Chain-Acyl CoA Dehydrogenase Deficiency
   * Trifunctional Protein Deficiency
   * Long Chain Hydroxyacyl-CoA Dehydrogenase Deficiency
   * Carnitine Palmitoyltransferase I or II Deficiency
   * Carnitine/Acylcarnitine Translocase Deficiency
   * Primary Carnitine Transport Deficiency
4. Hypoxic-Ischemic Encephalopathy

Exclusion Criteria:

* Prior Solid-Organ Transplant
* Use of any other investigational drug, biologic, or therapy or any clinical or laboratory abnormality or medical condition that, as determined by the investigator, may interfere with or obscure the biomarker measurements

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible subjects will be recruited from the patient population at Children's National Hospital in Washington, DC. Study population will consist of those patients with inherited hyperammonemias, acute metablic disorders, fatty acid oxidation disorders, and hypoxic-ischemic encephalopathy.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Biomarker Brain Injury Chronology | 2 Years
  Determine the chronology of biomarkers of brain injury (S100B, NSE, and UCHL1) in response to a hyperammonemic (HA) brain insult in patients with an inherited hyperammonemic disorder

SECONDARY OUTCOMES:
Brain Injury Protein Alterations | 2 Years
  Determine if S100B, NSE, and UCHL1 are altered in patients with two other inborn errors of metabolism in which the primary pathology is neurological injury, Maple Syrup Urine Disease (MSUD) and Glutaric Acidemia (GA1)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Ah Mew, MD, Principal Investigator — Children's National Research Institute; Ljubica Caldovic, PhD, Study Chair — Children's National Research Institute
Locations (1):
- Children's National Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided